CLINICAL TRIAL: NCT00921206
Title: Open-label Study to Investigate the Humoral and Cellular Immune Response to Two Doses of VAX102 Influenza Vaccine in Healthy Adults
Brief Title: Study to Investigate the Immune Response to Two Doses of VAX102 Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VaxInnate Corporation (Industry)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAX102-05
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Influenza
Keywords: influenza; influenza vaccine; universal influenza vaccine; Matrix 2e protein; M2e; Immune response
MeSH Terms: conditions — Influenza, Human | interventions — VAX102 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VAX102 given i.m. (Active Comparator): Universal influenza candidate vaccine
  Interventions: Biological: VAX102
- VAX102 given s.c. (Active Comparator): Universal influenza candidate vaccine
  Interventions: Biological: VAX102

INTERVENTIONS:
Biological: VAX102 — 1 ug i.m. compared to 2 ug s.c.
  Other Names: STF2.4xM2e

SUMMARY:
The objective is to assess the humoral and cellular immune response of the VAX102 vaccine delivered IM and SC in a prime-boost regimen at dose levels 1 µg or 2 µg in healthy adults against the influenza A virus M2e antigen after each vaccination.

DETAILED DESCRIPTION:
The primary objective is to assess the humoral and cellular immune response of the VAX102 vaccine delivered IM and SC in a prime-boost regimen at dose levels 1 µg or 2 µg in healthy adults against the influenza A virus M2e antigen after each vaccination. The magnitude and quality of the M2e-specific B and T cells will be measured. B cell responses will be evaluated on pre-dose Days 0, 28 and post-dose Days 7, 35, 42 and 60. T cell responses will be measured on pre-dose Days 0, 28 and post-dose Days 14, 42 and 60. IgG M2e antibody will be measured on Days 0, 7, 14, 28, 35. 42 and 60. The secondary objective is to assess the safety, reactogenicity, and tolerability of the VAX102 vaccine delivered IM or SC at dose levels 1 µg or 2 µg, in a prime-boost dosing regimen, in healthy adults 18-49 years of age, inclusive.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 - 49 years inclusive
* Give written informed consent to participate.
* Healthy, as determined by medical history, physical examination, vital signs, and clinical safety laboratory examinations
* Females willing to practice birth control to avoid pregnancy during the study
* Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits.

Exclusion Criteria:

* Presence of significant acute or chronic, uncontrolled medical or psychiatric illness (institution of new medical or surgical treatment, or a significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months) as determined by medical history and/or physical exam.
* Cancer, or treatment for cancer, within 3 years. Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible
* Impaired immune responsiveness (of any cause), including diabetes mellitus.
* Documented influenza infection in the 6 months prior to study entry.
* Presently receiving or history of receiving any medications or treatments that affects the immune system such as allergy shots, immune globulin, interferon, immunomodulators, cytotoxic drugs or drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable) in the past 6 months. Inhaled and topical corticosteroids will be allowed.
* Receipt or planned administration of a nonstudy vaccine within 30 days before and during the study and through the Day 42 evaluation.
* History of anaphylactic type reaction to injected vaccines.
* History of drug or chemical abuse in the year before the study.
* Use of new prescription medications started within 7 days before study entry.
* Receipt of blood or blood products 8 weeks before study entry or planned administration during the study period.
* Donation of blood or blood products within 8 weeks before study entry or at any time during the study.
* Acute disease within 72 hours prior to vaccinations, defined as the presence of a moderate or severe illness (as determined by the investigator through medical history and physical examination; for example, those requiring an absence from work) with or without fever, or a fever >37.9ºC orally. Study vaccine can be administered to persons with a minor illness, such as diarrhea, or mild upper respiratory tract infection with or without low-grade febrile illness. Vaccination can be delayed until the subject has recovered.
* Any condition that, in the opinion of the investigator, might interfere with study objectives

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2009-06; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To assess the humoral and cellular immune response of the VAX102 vaccine delivered IM and SC in a prime-boost regimen at dose levels 1 µg or 2 µg in healthy adults against the influenza A virus M2e antigen after each vaccination. | 2 months

SECONDARY OUTCOMES:
To assess the safety, reactogenicity, and tolerability of the VAX102 vaccine delivered IM or SC at dose levels 1 µg or 2 µg, in a prime-boost dosing regimen, in healthy adults 18-49 years of age, inclusive. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward Janoff, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Universite of Colorado, Denver, Denver, Colorado, United States

REFERENCES:
- See also: Sponsor website — http://www.vaxinnate.com/